CLINICAL TRIAL: NCT04400383
Title: An Open, Two-stage, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AB011 Injection in Patients With CLDN18.2-positive Advanced Solid Tumors
Brief Title: Clinical Trial to Evaluate AB011 Injection in Patients With CLDN18.2-positive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB011-ST-01
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor; Gastric Cancer; Pancreatic Adenocarcinoma
Keywords: advanced solid tumors; Gastric Cancer; Esophagogastric Junction Cancer; Pancreatic Adenocarcinoma; Claudin 18.2; CLDN18.2; monoclonal antibody
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AB011 Injection (Experimental): AB011 Injection treatment. This phase 1 trial will include two stages, a single treatment stage and a Combo treatment stage.
  Interventions: Drug: AB011 Injection

INTERVENTIONS:
Drug: AB011 Injection — Stage 1 Single treatment: AB011 Injection with dose escalation of 1mg/kg up to 40mg/kg, as well as dose expansion with recommended dose level from dose escalation.
  Stage 2 Combo Treatment: AB011 combine XELOX( GC) or Gem/nab-P (PC) Injection with dose escalation of 10mg/kg up to 30mg/kg, as well as dose expansion with recommended dose level from dose escalation.
  Other Names: recombinant humanized anti-Claudin 18.2 monoclonal antibody injection; recombinant humanized anti-CLDN 18.2 monoclonal antibody injection

SUMMARY:
This is an open, two-stage, phase I study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of AB011 injection in patients with CLDN18.2-positive advanced solid tumors.

DETAILED DESCRIPTION:
This study is an open, two-stage, phase I study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of AB011 injection in patients with CLDN18.2-positive advanced solid tumors. The study is composed of two stages: stage I is single treatment and stage II is combo treatment.

ELIGIBILITY:
Stage 1:

Inclusion Criteria:

* 1. Aged 18 to 80 years, either sex;
* 2. Patients with histologically or cytologic confirmed advanced solid tumors should have failed the standard treatment, or have no standard treatment regimen available, or have no access to standard treatment;
* 3. Tumor tissue samples is CLDN18.2 positive;
* 4. According to RECIST1.1, there are at least one evaluable tumor lesion during dose escalation period (stage 1), and at least one measurable tumor lesion during dose expansion period (stage 2);
* 5. The ECOG score is 0 to 1;
* 6. Expected survival > 3 months;
* 7. Various organs in good condition;
* 8. Fertile eligible patients (male and female) and their partners are willing to use a reliable method of contraception (hormones, barriers or abstinence) during the study and within 90 days after the last study treatment; women of childbearing potential must be tested for serum or urine pregnancy within 7 days before enrollment with negative results;
* 9. Patients are informed of this study before the trial and sign written informed consent form.

Exclusion Criteria:

* 1. Received anti-tumor therapies within 4 weeks prior to first administration of study drug, except: within 6 weeks for nitrosoureas or mitomycin C, within 2 weeks or 5 half-life of drugs (whichever longer) for oral fluorouracils and small molecular targeted drugs, and within 2 weeks for traditional Chinese medicines with indications of anti-tumor;
* 2. Received other non-marketed clinical trial drugs within 4 weeks prior to first administration of study drugs;
* 3. Received major surgery or had significant trauma within 4 weeks prior to first administration of study drug;
* 4. Received systemic corticosteroids or other immunosuppressors within 14 days prior to first administration of study drug;
* 5. Patients with AEs from previous treatment that have not recovered to ≤1 (CTCAE 5.0 );
* 6. Patients have central nervous system (CNS) metastasis or meningeal metastasis, or other evidences which demonstrate the CNS metastasis or meningeal metastasis are not controlled, resulting that patients are not eligible for enrollment at the investigator's discretion;
* 7. Patients with any active infection which requires systemic treatment with of anti-infection currently;
* 8. Patients with medical history of immune deficiency;
* 9. Patients with hepatitis B;
* 10.Patients with HCV infection but who with the HCV-RNA lower than the lower limit of detection can be enrolled ;
* 11.Patients with interstitial lung disease or Pulmonary function abnormalities which were identified by the investigator as clinically significant;
* 12.Patients who received any anti-CLDN18.2 treatment;
* 13.Patients with significant medical history of cardiovascular and cerebrovascular diseases;
* 14.Patient with high risks of gastrointestinal hemorrhage at the investigator's discretion;
* 15.Patients who need long-term use of non-steroidal anti-inflammatory drugs (NSAIDs) ;
* 16.Known alcohol use or drug dependence;
* 17.Patients with mental disorders or poor compliance;
* 18.Pregnant or lactating women;
* 19.Past severe allergic reactions or allergies to known components of AB011 injection ;
* 20.Persistent recurrent vomiting (defined as ≥3 vomiting in 24 hours);
* 21. Have other uncured malignant tumors in the past 5 years or at the same time, except cervical carcinoma in situ, basal cell carcinoma of the skin and other tumors with very low malignant degree;
* 22.Live attenuated vaccine was administered within 4 weeks prior to initial administration of the study drug;
* 23.Patients who with other serious systemic diseases or cannot participate in this trial due to other reasons, at the investigator's discretion.

Stage 2:

Inclusion Criteria:

* 1. Aged 18 to 80 years, either sex;
* 2. Patients with histologically or cytologic confirmed advanced gastric/oesophagus- gastric junction cancer or pancreatic cancer without systemic therapy (neoadjuvant therapy or postoperative adjuvant therapy, no tumor progression or recurrence within 6 months of last medication)
* 3. Tumor tissue samples is CLDN18.2 positive ;
* 4. According to RECIST1.1, there are at least one evaluable tumor lesion during dose escalation period (stage 1), and at least one measurable tumor lesion during dose expansion period (stage 2);
* 5. The ECOG score is 0 to 1;
* 6. Expected survival > 3 months;
* 7. Various organs in good condition;
* 8. Fertile eligible patients (male and female) and their partners are willing to use a reliable method of contraception (hormones, barriers or abstinence) during the study and within 90 days after the last study treatment; women of childbearing potential must be tested for serum or urine pregnancy within 7 days before enrollment with negative results;
* 9. Patients are informed of this study before the trial and sign written informed consent form.

Exclusion Criteria:

* 1. Received any other unmarketed investigational drug within 4 weeks prior to initial use of the investigational drug;
* 2. Patients with gastric adenocarcinoma and gastric cancer/esophagogastric junction adenocarcinoma have allergies, intolerations, contraindications or other unsuitable applications of capecitabine or oxaliplatin regimen (such as complete lack of known dihydropyrimidine dehydrogenase activity, etc.);Subjects with pancreatic cancer have allergies, intolerations, contraindications, or other inappropriate use of gemcitabine, other drugs or any of the components that may be used in the albumin-bound paclitaxel regimen;
* 3. If the patient has received local treatment such as radiotherapy for locally advanced unresectable or metastatic gastric/oesophagogastric junction cancer or pancreatic cancer, unless the treatment was completed >28 days before the first administration of the study drug.Patients who received palliative radiotherapy with peripheral bone metastases and recovered from all acute toxicity ≥ 14 days prior to initial administration of the study therapy were eligible for inclusion;
* 4. Patients with gastric/oesophagogastric junction carcinoma are known to have grade ≥2 peripheral sensory neuropathy, unless loss of deep tendon reflex is the only neurological abnormality;
* 5. Major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to initial use of the study drug;
* 6.Received systemic glucocorticoid (prednisone > 10mg/ day or equivalent dose of the same drug) or other immunosuppressant treatment within 14 days prior to initial use of the study drug; The exceptions are: local, ocular, intraarticular, intranasal, and inhaled glucocorticoids;Short-term use of glucocorticoids for prophylactic treatment (e.g. to prevent contrast allergy);
* 7.Patients with AEs from previous treatment that have not recovered to ≤1(CTCAE 5.0）;
* 8. Patients have central nervous system (CNS) metastasis or meningeal metastasis, or other evidences which demonstrate the CNS metastasis or meningeal metastasis are not controlled, resulting that patients are not eligible for enrollment at the investigator's discretion;
* 9. Patients with any active infection which requires systemic treatment with of anti-infection currently;
* 10. Patients with medical history of immune deficiency, Including positive HIV antibodies;
* 11. Patients with hepatitis B;
* 12.Patients with HCV infection but who with the HCV-RNA lower than the lower limit of detection can be enrolled ;
* 13.Patients who have interstitial lung disease or Pulmonary function abnormalities which were identified by the investigator as clinically significant;
* 14.Patients received any anti-CLDN18.2 treatment;
* 15.Patients with have significant medical history of cardiovascular and cerebrovascular diseases;
* 16.Patient with high risks of gastrointestinal hemorrhage at the investigator's discretion;
* 17.Patients who need long-term use of non-steroidal anti-inflammatory drugs (NSAIDs) ;
* 18.Known alcohol use or drug dependence;
* 19.Patients with mental disorders or poor compliance;
* 20.Pregnant or lactating women;
* 21.Past severe allergic reactions or allergies to known components of AB011 injection;
* 22.Persistent recurrent vomiting (defined as ≥3 vomiting in 24 hours);
* 23. Have other uncured malignant tumors in the past 5 years or at the same time, except cervical carcinoma in situ, basal cell carcinoma of the skin and other tumors with very low malignant degree;
* 24.Live attenuated vaccine was administered within 4 weeks prior to initial administration of the study drug;
* 25.Patients have other serious systemic diseases or cannot participate in this trial due to other reasons, at the investigator's discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Stage1：Incidence of adverse events AE of single and multiple dose (according to NCI CTCAE 5.0) | From First dose to last patient progression or 6 months, whichever came first
  An AE or SAE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Stage1：Incidence of adverse events SAE of single and multiple dose (according to NCI CTCAE 5.0) | From First dose to last patient progression or 6 months, whichever came first
  An AE or SAE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Stage 1: The incidence and case number of DLT (Dose Limiting Toxicity) during observation period | From first dose up to 28 days
  DLT is short for Dose Limiting Toxicity. dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Stage 2：Incidence of adverse events AE of single and multiple dose for AB011 combinate with XELOX or Gem/nab-P (according to NCI CTCAE 5.0) | From First dose to last patient progression or 12 months, whichever came first
  An AE or SAE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Stage 2：Incidence of adverse events SAE of single and multiple dose for AB011 combinate with XELOX or Gem/nab-P (according to NCI CTCAE 5.0) | From First dose to last patient progression or 12 months, whichever came first
  An AE or SAE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Stage 2: The incidence and case number of DLT (Dose Limiting Toxicity) during observation period | From first dose up to 21 days
  DLT is short for Dose Limiting Toxicity. dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.

SECONDARY OUTCOMES:
Stage 1: Pharmacokinetics: Area Under Curve (AUC) with immunoanalytical method | Up to progression of disease after injection, or end of 6 cycle( each cycle is 28 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: Pharmacokinetics: Area Under Curve (AUC) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 1: Pharmacokinetics: clearance rate (CL) with immunoanalytical method | Up to progression of disease after injection, or 6 cycle( dose increase), 8 cycle (dose extension), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: Pharmacokinetics: clearance rate (CL) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 1: Pharmacokinetics: minimum concentration (Cmin) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6（dose increase stage), or cycle 8 (dose expansion stage), each cycle is 28 days, whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: Pharmacokinetics: minimum concentration (Cmin) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 1: Pharmacokinetics: maximum concentration (Cmax) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6（dose increase stage), or cycle 8 (dose expansion stage), each cycle is 28 days, whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: Pharmacokinetics: maximum concentration (Cmax) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 1: Pharmacokinetics: half-life (T1/2) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6（dose increase stage), or cycle 8 (dose expansion stage), each cycle is 28 days, whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: Pharmacokinetics: half-life (T1/2) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 1: volume of distribution (Vd) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6（dose increase stage), or cycle 8 (dose expansion stage), each cycle is 28 days, whichever came first
  AUC will be recorded from the PK serum samples collected.
Stage 2: volume of distribution (Vd) with immunoanalytical method | Up to progression of disease after injection, or end of cycle 6 (each cycle is 21 days), whichever came first
  AUC will be recorded from the PK serum samples collected.
Immunogenicity | Up to 8 months (end of treatment)
  Incidence of anti-drug antibodies
Efficacy: objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to progression of disease after injection, or 6 months( stage 1), 12 months (stage 2) whichever came first
  These measure are defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
Efficacy: disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to progression of disease after injection, or 6 months( stage 1), 12 months (stage 2) whichever came first
  These measure are defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
Efficacy: duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to progression of disease after injection, or 6 months( stage 1), 12 months (stage 2) whichever came first
  These measure are defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
Efficacy: progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to progression of disease after injection, or 6 months( stage 1), 12 months (stage 2) whichever came first
  These measure are defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
Efficacy: overall survival (OS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to progression of disease after injection, or 6 months( stage 1), 12 months (stage 2) whichever came first
  These measure are defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital
Locations (12):
- China (12):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Huaihua Second People's Hospital, Huaihua, Hunan
  - Linyi Cancer Hospital, Linyi, Shandong
  - Zhongshan Hospital, Zhongshan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No